CLINICAL TRIAL: NCT06388655
Title: The Effect of the Mobile EEG-Neurofeedback in Healthy Child and Adolescent Participants: a Randomized Sham-control Study
Brief Title: The Effect of the Mobile EEG-Neurofeedback in Healthy Child and Adolescent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Junwon Kim, Clinical professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MDCR-19-007
Record Dates: First submitted 2024-04-15; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Internet Addiction
Keywords: mobile neurofeedback; neurotypical; internet addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MNF active group (Experimental): In this study, neurofeedback headsets developed by OmniCNS were utilized, employing a dry EEG method to measure EEG signals at a rate of 250Hz. Signals were then transformed into the frequency domain through Fourier transform, allowing assessment of power across a wide range of frequencies. Feedback activities, like levitation or running, were based on attention levels determined by the Low beta + Middle beta / Theta Power ratio. Participants received training and engaged in neurofeedback games through the Omnifit Brain app using the provided headsets and personal smartphones for 12 weeks, three times a week for 10-20 minutes per session. Four game types based on the theta/beta ratio were offered, allowing participants to choose freely.
  Interventions: Device: mobile neurofeedback
- sham control group (Sham Comparator): The sham neurofeedback was implemented through presenting randomized game outcomes, independent of real measurements. The scoring distribution was meticulously adjusted to achieve a realistic spectrum of results, prioritizing median scores to uphold uniformity in user experience.
  Interventions: Device: sham mobile neurofeedback

INTERVENTIONS:
Device: mobile neurofeedback — The participants were randomly assigned to the MNF active (N=31) or sham control (N=30) groups. The MNF program was administered using a mobile app (equipped with a headset with a 2-channel EEG sensor) for 30 min/day, 3 days/week, for 3 months.
  Arms: MNF active group
Device: sham mobile neurofeedback — The sham neurofeedback was implemented through presenting randomized game outcomes, independent of real measurements. The scoring distribution was meticulously adjusted to achieve a realistic spectrum of results, prioritizing median scores to uphold uniformity in user experience.
  Arms: sham control group

SUMMARY:
The objective of this study was to ascertain the therapeutic impact of mobile neurofeedback (MNF) in neurotypical children when compared to sham MNF. Clinical assessments were conducted both before and after the MNF intervention, and the effectiveness of the intervention was to be validated through these evaluations.

DETAILED DESCRIPTION:
Neurotypical children aged 10-15 participated in the study. All subjects were assessed using the Kiddie Schedule for Affective Disorders and Schizophrenia Present and Lifetime Version Korean Version (K-SADS-PL-K) and confirmed to have no psychiatric symptoms. The participants were randomly assigned to the MNF active (N=31) or sham control (N=30) groups. The MNF program was administered using a mobile app (equipped with a headset with a 2-channel EEG sensor) for 30 min/day, 3 days/week, for 3 months. All participants and their parents completed self-report scales and participants complete neurocognitive function assessments including the continuous performance test, Stroop, children's color trails test-1 and 2, and intelligence test at baseline and after the 3-month MNF program.

ELIGIBILITY:
Inclusion Criteria:

Child participants ranging from 8 to 15 years of age, who were recruited from the Department of Psychiatry at Daegu Catholic University Medical Center between 2019 and 2021

Exclusion Criteria:

History of congenital genetic diseases History of brain damage History of neurological disorders History of psychiatric conditions such as schizophrenia spectrum disorder, autism spectrum disorder, obsessive-compulsive disorder, major depressive disorder, or bipolar disorder Participants with an IQ below 70, as determined by the Korean-Wechsler Intelligence Scale for Children-Fourth Edition (K-WISC-IV)

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Comparisons of the means of children's self-scale variables | through study completion, an average of 1 year
  Participants' condition regarding internet addiction, among other factors, was assessed using children's self-scales such as the Korea Internet Addiction Scale (K-scale).

SECONDARY OUTCOMES:
Comparisons of the means of parents' self-scale variables : Beck Depression Inventory-II (BDI-II) | through study completion, an average of 1 year
  The evaluation of participants was conducted using parents' self-scales : Beck Depression Inventory-II (BDI-II)
Comparisons of the means of parents' self-scale variables : Beck Anxiety Inventory (BAI) | through study completion, an average of 1 year
  The evaluation of participants was conducted using parents' self-scales : Beck Anxiety Inventory (BAI)
Comparisons of the means of children's K-WISC-IV(Korean Wechsler Intelligence Scale for Children-IV) | through study completion, an average of 1 year
  Participants' intelligence levels were assessed using measures
Comparisons of the means of children's Stroop | through study completion, an average of 1 year
  Participants' attention levels were assessed using measures
Comparisons of the means of children's ATA(Advanced Test of Attention) | through study completion, an average of 1 year
  Participants' attention levels were assessed using measures
Comparisons of the means of children's CCTT(Children's Color Trails Test) | through study completion, an average of 1 year
  Participants' attention levels were assessed using measures

CONTACTS AND LOCATIONS:
Locations (1):
- Daegu Catholic University Medical Center, Daegu, Nam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No